CLINICAL TRIAL: NCT07273084
Title: Multidisciplinary Intervention in Patients With Non-Cancer Chronic Pain in a Primary Care Center: Pilot Study
Brief Title: Multidisciplinary Intervention for Non-Cancer Chronic Pain: Pilot Study
Acronym: MICNP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Victor Ortiz Mallasen (Other)
Responsible Party: Sponsor-Investigator, Victor Ortiz Mallasen, Assistant Professor of Nursing, Universitat Jaume I
Organization: Universitat Jaume I (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PILOT-12PAT-2025
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non-cancer Pain; Chronic Non-cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Multidisciplinary Intervention (Experimental): All participants will receive a multidisciplinary intervention program lasting 6 weeks, consisting of 17 sessions that combine pain neuroscience education, individualized therapeutic exercises, and promotion of healthy lifestyle habits. The program aims to improve pain management skills and health-related quality of life in patients with non-cancer chronic pain.
  Interventions: Behavioral: Multidisciplinary Intervention Program for Chronic Non-Cancer Pain

INTERVENTIONS:
Behavioral: Multidisciplinary Intervention Program for Chronic Non-Cancer Pain — A 6-week multidisciplinary group program composed of 17 sessions combining pain neuroscience education, individualized therapeutic exercises, and promotion of healthy lifestyle habits. The intervention aims to improve pain management skills, physical function, and health-related quality of life in adults with non-cancer chronic pain.

SUMMARY:
Introduction:

Non-cancer chronic pain (NCCP) persists beyond the injury that caused it, affecting approximately 20% of the global population (around 1.6 billion people) and 17-18% in Spain (about 8 million people). Its treatment is complex and often insufficient, highlighting the need for an integrated, multimodal, multidisciplinary approach coordinated between primary and hospital care.

Objective:

To evaluate the effectiveness of a multidisciplinary intervention program combining pain neuroscience education, therapeutic physical exercise, and promotion of healthy habits, aiming to improve health-related quality of life in individuals with NCCP at the Benicàssim Health Center.

Methodology:

This is a quasi-experimental, before-and-after pilot study, non-randomized, without a control group, using a convenience sample of 12 participants. Sociodemographic, health-related, and clinical variables will be measured, including health-related quality of life, central sensitization, kinesiophobia, catastrophizing, pain level, body mass index, sleep quality, perceived social support, anxiety, and depression. Measurements will be taken before the program, at completion, and at 3 months.

The intervention is a 6-week group program with 17 sessions, combining pain neuroscience education, individualized therapeutic exercises, and promotion of healthy habits. Data will be analyzed using SPSS v.29 with a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 79 years.
* Individuals diagnosed with non-cancer chronic pain lasting more than 3 months.

Exclusion Criteria:

* Individuals with pain of oncologic origin.
* Individuals who have experienced a fracture or undergone surgery within the past year.
* Pregnant women.
* Individuals without adequate understanding of the Spanish language.
* Individuals with cognitive impairment that prevents them from performing the program's interventions.
* Individuals with physical performance deficits that prevent them from carrying out the program's activities.
* Individuals with urinary and/or fecal incontinence.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life Measured With the EQ-5D-5L | Baseline, immediately after the 6-week program, and 3 months after intervention completion.
  Health-related quality of life will be assessed using the EQ-5D-5L questionnaire. The EQ-5D-5L index value typically ranges from less than 0 (worse than death) to 1.00 (full health). Higher scores indicate better health-related quality of life. The EQ-VAS ranges from 0 (worst imaginable health) to 100 (best imaginable health).

SECONDARY OUTCOMES:
Pain Intensity Measured With the Visual Analog Scale (VAS) | Baseline, post-intervention, 3 months.
  Pain intensity will be measured using the Visual Analog Scale (VAS), a 100-mm line ranging from 0 (no pain) to 100 (worst imaginable pain). Higher scores indicate worse pain intensity.
Central Sensitization Assessed With the Central Sensitization Inventory (CSI) | Baseline, immediately after the intervention, and 3 months after intervention completion.
  Central sensitization will be assessed using the Central Sensitization Inventory (CSI), consisting of 25 items scored from 0 to 4. The total score ranges from 0 (no symptoms) to 100 (maximum symptom severity). Higher scores indicate worse central sensitization.
Kinesiophobia Measured With the Tampa Scale for Kinesiophobia (TSK-11) | Baseline, immediately after the intervention, and 3 months after intervention completion.
  Fear of movement will be assessed using the 11-item Tampa Scale for Kinesiophobia (TSK-11). Scores range from 11 (lowest fear) to 44 (highest fear). Higher scores indicate worse kinesiophobia.
Pain Catastrophizing Measured With the Pain Catastrophizing Scale (PCS) | Baseline, immediately after the intervention, and 3 months after intervention completion.
  Pain catastrophizing will be measured using the Pain Catastrophizing Scale (PCS), a 13-item questionnaire. Scores range from 0 (no catastrophizing) to 52 (maximum catastrophizing). Higher scores indicate worse catastrophizing.
Sleep Quality Assessed With the Pittsburgh Sleep Quality Index (PSQI) | Baseline, immediately after the intervention, and 3 months after intervention completion.
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The global score ranges from 0 (better sleep quality) to 21 (poorer sleep quality). Higher scores indicate worse sleep quality.
Anxiety and Depression Assessed With the Hospital Anxiety and Depression Scale (HADS) | Baseline, immediately after the intervention, and 3 months after intervention completion.
  Anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS), which includes two subscales (anxiety and depression), each ranging from 0 (no symptoms) to 21 (severe symptoms). Higher scores indicate worse anxiety or depression.
Perceived Social Support Measured With the Duke-UNC Functional Social Support Questionnaire | Baseline, immediately after the intervention, and 3 months after intervention completion.
  Perceived social support will be assessed using the Duke-UNC Functional Social Support Questionnaire. Scores range from 8 (lowest support) to 40 (highest support). Higher scores indicate better perceived social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Benicassim Health Center, Benicassim, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No